CLINICAL TRIAL: NCT01662492
Title: 191622-103 BOTOX® (Botulinum Toxin Type A) Purified Neurotoxin Complex as Headache Prophylaxis in Adolescents (Children 12 to < 18 Years of Age) With Chronic Migraine
Brief Title: A Study Using Botulinum Toxin Type A as Headache Prophylaxis in Adolescents With Chronic Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 191622-103
Record Dates: First submitted 2012-08-08; First posted 2012-08-10 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-07

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Botulinum toxin type A Dose 1 (Experimental): Botulinum toxin type A Dose 1 intramuscular injections into specified muscles.
  Interventions: Biological: Botulinum toxin type A Dose 1
- Botulinum toxin type A Dose 2 (Experimental): Botulinum toxin type A Dose 2 intramuscular injections into specified muscles.
  Interventions: Biological: Botulinum toxin type A Dose 2
- Placebo (Normal Saline) (Placebo Comparator): Placebo (Normal Saline) intramuscular injections into specified muscles.
  Interventions: Drug: Placebo (Normal Saline)

INTERVENTIONS:
Biological: Botulinum toxin type A Dose 1 — Botulinum toxin type A Dose 1 intramuscular injections into specified muscles.
  Other Names: onabotulinumtoxinA; BOTOX®
  Arms: Botulinum toxin type A Dose 1
Biological: Botulinum toxin type A Dose 2 — Botulinum toxin type A Dose 2 intramuscular injections into specified muscles.
  Other Names: onabotulinumtoxinA; BOTOX®
  Arms: Botulinum toxin type A Dose 2
Drug: Placebo (Normal Saline) — Placebo (Normal Saline) intramuscular injections into specified muscles.
  Arms: Placebo (Normal Saline)

SUMMARY:
To evaluate the efficacy and safety of Botulinum Toxin Type A versus placebo (normal saline) as headache prophylaxis in adolescents (children 12 to 17) with chronic migraine.

ELIGIBILITY:
Inclusion Criteria:

* Medical history of chronic migraine for at least 6 months
* 15 or more headache days during a 4 week period

Exclusion Criteria:

* Previous use of any botulinum toxin of any serotype for any reason
* Diagnosis of Myasthenia gravis, Eaton-Lambert Syndrome, Amyotrophic Lateral Sclerosis
* Treatment of headache using acupuncture, transcutaneous electrical stimulation (TENS), cranial traction, dental splints, or injection of anesthetics/steroids within 4 weeks prior to the week -4 screening visit
* Use of any headache prophylaxis medication within 4 weeks prior to the week -4 screening visit

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2012-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (22):
- United States (22):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Fullerton Neurology and Headache Center, Fullerton, California
  - The Research Center of Southern California, Oceanside, California
  - San Francisco Clinical Research Center, San Francisco, California
  - Stanford Hospital and Clinics, Stanford, California
  - Associated Neurologists of Southern CT, P.C., Fairfield, Connecticut
  - New England Institute for Clinical Research, Stamford, Connecticut
  - NW FL Clinical Research Group, LLC, Gulf Breeze, Florida
  - Pediatric Neurology, PA, Orlando, Florida
  - The Premiere Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - Advanced Clinical Research, Meridian, Idaho
  - Josephson Wallack Munshower Neurology, P.C., Indianapolis, Indiana
  - CPFCC Neurology Research Department, Overland Park, Kansas
  - Michigan Head Pain & Neurological Institute, Ann Arbor, Michigan
  - CORE (Center for Outpatient Research), Springfield, Missouri
  - Renown Institution for Neurosciences, Reno, Nevada
  - Rochester Clinical Research, Inc, Rochester, New York
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Jill Waldo, CCRC, Pittsburgh, Pennsylvania
  - Nashville Neuroscience Group, Nashville, Tennessee
  - Texas Association of Pediatric Neurology/Road Runner Research, San Antonio, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah

REFERENCES:
- [Derived] Shah S, Calderon MD, Wu W, Grant J, Rinehart J. Onabotulinumtoxin A (BOTOX(R)) for ProphylaCTIC Treatment of Pediatric Migraine: A Retrospective Longitudinal Analysis. J Child Neurol. 2018 Aug;33(9):580-586. doi: 10.1177/0883073818776142. Epub 2018 Jun 7. PMID 29877131
- See also: More Information — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Botulinum Toxin Type A 155 U: Botulinum toxin type A, 155 U, intramuscular injections into specified muscles.
- Botulinum Toxin Type A 74 U: Botulinum toxin type A, 74 U, intramuscular injections into specified muscles.
Period: Overall Study
Arm/Group | Botulinum Toxin Type A 155 U | Botulinum Toxin Type A 74 U | Placebo (Normal Saline)
Started | 45 | 43 | 37
Completed | 42 | 42 | 31
Not Completed | 3 | 1 | 6
Not completed — Other miscellaneous reasons. | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Lack of Efficacy | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A 155 U | Botulinum Toxin Type A 74 U | Placebo (Normal Saline) | Total
Number analyzed (Participants) | 45 | 43 | 37 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.1 (1.4) | 15.0 (1.5) | 15.2 (1.5) | 15.1 (1.5)
Sex/Gender, Customized [Number; unit: participants]
  Male | 8 | 11 | 8 | 27
  Female | 37 | 32 | 29 | 98

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Frequency of Headache Days
Description: Change from baseline in the frequency of headache days during the 28-day period, ending with Week 12 in the Intent-to-Treat population. A headache day for a patient is defined as a calendar day with 1 or more total hours of headache as recorded by the patient in the electronic diary.
Time Frame: Baseline, 12 Weeks
Population: Intent-to-Treat (ITT) Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: Headache days
Arm/Group | Botulinum Toxin Type A 155 U | Botulinum Toxin Type A 74 U | Placebo (Normal Saline)
Number analyzed (Participants) | 45 | 43 | 37
Headache days
  Baseline | 23.2 (4.4) | 23.4 (4.8) | 25.3 (3.9)
  Change from Baseline at Week 12 | -6.3 (7.0) | -6.4 (7.8) | -6.8 (8.2)

2. Secondary Outcome: Change From Baseline in the Frequency of Severe Headache Days
Description: Change from baseline in the frequency of severe headache days during the 28-day period, ending with Week 12 in the Intent-to-Treat population. A severe headache day is defined as a calendar day with 1 or more total hours of headache and with maximum severity reported as 'severe' for the day as recorded by the patient in the electronic diary.
Time Frame: Baseline, 12 Weeks
Population: Intent-to-Treat (ITT) Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: Severe Headache Days
Arm/Group | Botulinum Toxin Type A 155 U | Botulinum Toxin Type A 74 U | Placebo (Normal Saline)
Number analyzed (Participants) | 45 | 43 | 37
Severe Headache Days
  Baseline | 7.0 (5.0) | 7.8 (6.2) | 9.1 (8.3)
  Change from Baseline at Week 12 | -1.3 (4.7) | -2.3 (6.3) | -0.9 (7.4)

3. Secondary Outcome: Change From Baseline in the Total Cumulative Hours of Headache on Headache Days
Description: Change From Baseline in the Total Cumulative Hours of Headache on Headache Days during the 28-day period ending with Week 12 in the Intent-to-Treat Population. Total cumulative hours is defined as the sum of total duration of headaches on headache days.
Time Frame: Baseline, 12 Weeks
Population: Intent-to-Treat (ITT) Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: Cumulative hours of headache
Arm/Group | Botulinum Toxin Type A 155 U | Botulinum Toxin Type A 74 U | Placebo (Normal Saline)
Number analyzed (Participants) | 45 | 43 | 37
Cumulative hours of headache
  Baseline | 170.69 (151.60) | 175.98 (139.76) | 212.68 (184.37)
  Change from Baseline at Week 12 | -36.52 (53.19) | -19.03 (113.73) | -50.04 (87.36)

4. Secondary Outcome: Percentage of Patients With ≥ 50% Decrease From Baseline in the Frequency of Headache Days
Description: Percentage of patients with ≥ 50% decrease from baseline in the frequency of headache days during the 28-day period ending with Week 12 in the Intent-to-Treat Population. A responder for headache days was defined as a patient with a 50% decrease in change from baseline in the frequency of headache days.
Time Frame: Baseline, 12 Weeks
Population: Intent-to-Treat (ITT) Population: All randomized subjects.
Measure: Number; unit: Percentage of participants
Arm/Group | Botulinum Toxin Type A 155 U | Botulinum Toxin Type A 74 U | Placebo (Normal Saline)
Number analyzed (Participants) | 45 | 43 | 37
Percentage of participants | 28.9 | 32.6 | 29.7

5. Secondary Outcome: Percentage of Patients Who Are Prescribed Oral Rescue Migraine Prophylactic Treatment
Description: Percentage of patients who are prescribed oral rescue migraine prophylactic treatment during the 28-day period ending with Week 12 in the Intent-to-Treat population.
Time Frame: 12 Weeks
Population: Intent-to-Treat (ITT) Population: All randomized subjects.
Measure: Number; unit: Percentage of participants
Arm/Group | Botulinum Toxin Type A 155 U | Botulinum Toxin Type A 74 U | Placebo (Normal Saline)
Number analyzed (Participants) | 45 | 43 | 37
Percentage of participants
  Week 4 | 0 | 0 | 0
  Week 8 | 4.4 | 9.3 | 2.7
  Week 12 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 12
Arm/Group | Botulinum Toxin Type A 155 U | Botulinum Toxin Type A 74 U | Placebo (Normal Saline)
Serious Adverse Events (participants affected / at risk) | 1/43 | 2/43 | 0/37
Other Adverse Events (participants affected / at risk) | 8/43 | 14/43 | 8/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A 155 U (N=43) | Botulinum Toxin Type A 74 U (N=43) | Placebo (Normal Saline) (N=37)
Cellulitis (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A 155 U (N=43) | Botulinum Toxin Type A 74 U (N=43) | Placebo (Normal Saline) (N=37)
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 3 | 4
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 1
Migraine (Nervous system disorders) | 1 | 3 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.